CLINICAL TRIAL: NCT03294655
Title: A Resilience Building Intervention to Promote Successful Aging
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pariya L. Fazeli, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Wheeler SON DSA
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Community Dwelling Adults Aged 50 and Older

STUDY DESIGN:
Intervention Model Description: pre-post experimental design, 60 adults aged 50+ will be randomized to either a no-contact control or intervention condition
Who Masked: Outcomes Assessor
Masking Description: only the post test assessor will be blinded to condition, as participants will know which condition they are assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No contact control (No Intervention): the no contact control group will do nothing
- Intervention (Experimental): the intervention condition will come to the lab for a 1 hour Pilot Resilience Building Intervention including a presentation on resilience and strategies to boost adherence, of which they will chose five to integrate in their daily life over the following 4 weeks
  Interventions: Behavioral: Pilot Resilience Building Intervention

INTERVENTIONS:
Behavioral: Pilot Resilience Building Intervention — The intervention will include a brief one-on-one visit in which psychoeducational information on building resilience will be given via a PowerPoint presentation, which will include exercises for the participants to engage in over the following four weeks in their daily lives. After the presentation participants will also develop a personalized intervention plan where they will choose at least five areas of the American Psychological Association 10 Strategies for Building Resilience on which to specifically focus. Participants will also receive a pamphlet of abbreviated information from the PowerPoint presentation.
  Arms: Intervention

SUMMARY:
In this pilot study, a pre-post experimental design will be used, in which 60 community dwelling adults aged 50+ will recruited from a larger parent study, and will then be randomized to either a no-contact control or intervention condition. Those in the intervention condition will receive a psychoeducational intervention in which they will receive scientific literature-based information on resilience and strategies to bolster resilience, as well as developing an individualized plan on areas to engage in at home over the next four weeks. All participants will return for an immediate posttest using an abbreviated version of the baseline battery from the parent study.

ELIGIBILITY:
Inclusion Criteria/Exclusion Criteria:

* Must be enrolled in a larger parent study
* The criteria for the parent study are: no neurological or severe neuromedical disorders (e.g., stroke, schizophrenia), must be able to speak English, not be legally blind or deaf, not currently undergoing chemotherapy or radiation therapy, no brain trauma with loss of consciousness greater than 30 mins, and not homeless.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Resilience | 4 weeks
  Connor Davidson Resilience Scale

CONTACTS AND LOCATIONS:
Locations (1):
- the Holly Mears Building/Center for Research on Applied Gerontology, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No